CLINICAL TRIAL: NCT05994378
Title: To Compare the Efficacy and Safety of Oral SHR7280 Tablets With Ganirelix Acetate Injection in Female Subjects With Infertility Receiving Controlled Ovarian Hyperstimulation Therapy: A Multi-center, Randomized, Parallel-Group, Double-Blind, Dual-Simulation, Non-Inferiority Phase III Clinical Study
Brief Title: To Compare the Efficacy and Safety of Oral SHR 7280 Tablets With Ganirelix Acetate Injection in Infertile Female Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR7280-302
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Infertile Female Subjects Undergoing Controlled Ovarian Hyperstimulation to Suppress Premature LH Surge and Prevent Early Ovulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: SHR7280；Ganirelix Acetate Injection simulant
- Control group (Active Comparator)
  Interventions: Drug: SHR7280 simulant； Ganirelix Acetate Injection

INTERVENTIONS:
Drug: SHR7280；Ganirelix Acetate Injection simulant — SHR7280 200mg Q12h and Ganirelix Acetate Injection simulant 0.5mL qd;
  Arms: Experimental group
Drug: SHR7280 simulant； Ganirelix Acetate Injection — SHR7280 simulant 200mg Q12h and Ganirelix Acetate Injection 0.5mL:0.25mg qd;
  Arms: Control group

SUMMARY:
This study is a multi-center, randomized, double-blind, positive drug-controlled, non-inferiority Phase III clinical trial. The study will enroll approximately 316 infertile female subjects undergoing controlled ovarian hyperstimulation (COH) for in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Married infertile female subjects aged 20 to 39 years with indications for in vitro fertilization-embryo transfer (IVF-ET) or intracytoplasmic sperm injection (ICSI);
2. Body mass index (BMI) 18 ~ 28kg/m2 (both exclusive) and weight 45Kg ~ 75Kg (both inclusive);
3. Regular menstrual cycle (24 ~ 35 days, both inclusive) for the last 3 months prior to screening;
4. Anticipated normal ovarian response;
5. Willingness of the subject to undergo fresh cycle transfer with one or two embryos at a time in the first IVF-ET cycle；
6. Normal cervical cytology results (TCT) or with limited clinically significance within 1 year prior to screening or on the screening visit; or subjects with atypical squamous cells of undetermined significance (ASC-US) of TCT tested negative for high-risk types of human papillomavirus (HPV);
7. Informed consent of subjects and their spouses;

Exclusion Criteria:

1. Prior to screening, individuals underwent three or more IVF/ICSI-ET COH cycles without achieving clinical pregnancy；
2. Previous IVF/ ICSI failure due to sperm/fertilization problems and no improvement in related medical condition;
3. Subjects with more than 2 times of spontaneous abortion;
4. Subjects at high risk of OHSS, judged by the investigator according to the Golan classification (e.g., those with moderate to severe OHSS during previous COH cycles, polycystic ovary syndrome (PCOS), or with previous cancelled COH cycles due to OHSS);
5. Subjects with decreased ovarian reserve;
6. TSH test result above or equal to 2.5 mIU/L for subjects with prior hypothyroidism or subclinical hypothyroidism on screening visit;
7. Any pregnancy that occurred within 3 months prior to screening visit;
8. Unexplained abnormal vaginal bleeding;
9. Infectious disease screening indicates any of the following: positive for HIV antibodies, positive for syphilis spirochete antibodies; positive for Hepatitis C virus (HCV) antibodies and positive HCV-RNA test; positive for Hepatitis B surface antigen (HBsAg) and HBV-DNA ≥ 1×103 kIU/L (or IU/mL);
10. Use of fertility regulators within one month before ovarian stimulation, such as clomiphene citrate, letrozole, gonadotropins (Gn), metformin, hormonal drugs (including oral contraceptives, estrogens, progestogens, etc.).
11. Past medical history or gynecological ultrasound indicates clinically significant conditions;
12. ALT and AST levels at the screening visit or the start of ovarian stimulation were more than twice the upper limit of normal;
13. Positive serum β-hCG test results on the screening visit or the start day of ovarian stimulation;
14. Blood or blood component donation within one month before screening, or a blood loss equivalent to at least 200 mL, or a blood transfusion within two months;
15. Severe infection, severe trauma, or major surgery within six months before screening;
16. Any disease or symptom that can affect systemic function and may affect the absorption, accumulation, metabolism, or excretion of the test drug (e.g., chronic intestinal diseases, Crohn's disease, ulcerative colitis).
17. Major systemic diseases, endocrine or metabolic abnormalities;
18. Thromboembolic diseases or a history of thromboembolic diseases;
19. The subject or her spouse requires oocyte or sperm donation, or either or both of them carry a chromosomal abnormality deemed clinically significant by the researcher, or suffer from a known monogenic hereditary disease or a severe disease with genetic susceptibility requiring pre-implantation genetic testing (PGT);
20. Smoking (more than 5 cigarettes or equivalent tobacco daily) or alcohol abuse (drinking ≥14 units of alcohol weekly: 1 unit = 360 mL beer, or 25 mL of 40% or higher spirits, or 1 glass of wine, 180 mL) within three months before screening;
21. History of drug abuse or drug dependence;
22. Allergic constitution or allergy to two or more foods or drugs, including a known allergy to any component of the test drug or non-test drug; contraindication or allergy to GnRH agonists or GnRH antagonists, recombinant or urinary FSH, hCG, progesterone drugs;
23. Participation in any drug or medical device clinical trial within three months before screening, or still in the follow-up period of a clinical study before screening, or within the 5 half-lives of the test drug (whichever is longer);
24. Malignant tumor or history of malignant tumor (except basal cell or squamous cell skin cancer, in situ cancer), or a high risk of malignant tumor onset/recurrence;
25. Known history of severe mental illness, or inability to understand the purpose, methods, etc., of this clinical trial, or non-compliance with research procedures;
26. Any other reasons deemed by the researcher as unsuitable for participation in this study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 317 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Number of oocyte retrieved per COH cycle | On oocyte retrieval 1 day
  number of oocytes obtained after one COH cycle;
Inhibition rate of premature LH surge | the hCG injection 1 day
  premature LH surge is defined as: LH ≥ 10 IU/L and progesterone P ≥ 1 ng/mL (3.18 nmol/L);

SECONDARY OUTCOMES:
2PN rate | 16-18 hours (h) after fertilization
  number of 2 pronuclei(2PN) oocytes/ number of oocytes retrieved or number of MII oocytes×100%;
High quality embryo rate | 3 days after fertilization
  number of high-quality embryos/ cleavage number×100%;
Chemical pregnancy rate | on chemical pregnancy test 1 day
  number of pregnancy cycles/ number of transplantation cycles×100%;
Clinical pregnancy rate | on clinical pregnancy test 1 day
  number of clinical pregnancy cycles/ number of transplantation cycles×100%;
Persistent pregnancy rate | on persistent pregnancy test 1 day
  number of clinical pregnancy cycles/ number of transplantation cycles×100%;
Adverse drug events | Day 1 to persistent pregnancy test day/ or End-of-trial visit 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided